CLINICAL TRIAL: NCT03797391
Title: First-in-human, Phase I/II, Multicenter, Open-Label Study of EMB-01 in Patients With Advanced/Metastatic Solid Tumors
Brief Title: A Dose Escalation With Expansion Study of EMB-01 in Participants With Advanced/Metastatic Solid Tumors
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai EpimAb Biotherapeutics Co., Ltd. (Industry)
Collaborators: Covance (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: EMB01X101
Record Dates: First submitted 2018-12-26; First posted 2019-01-09 (Actual); Last update posted 2023-05-31 (Actual); Status verified 2023-05

CONDITIONS: Neoplasms; Neoplasm Metastasis; Non-Small-Cell Lung Cancer
Keywords: Human Bispecific antibody,; Epidermal Growth Factor Receptor (EGFR),; c-Mesenchymal-Epithelial Transition (cMet),; Neoplasms, Neoplasm Metastasis,; Non-Small-Cell Lung Cancer (NSCLC), First-in-human,; EMB-01, Tyrosine Kinase Inhibitor (TKI) Resistant
MeSH Terms: conditions — Neoplasms; Neoplasm Metastasis; Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Intervention Model Description: Dose escalation followed by Protocol at 100mg, 200mg, 350mg, 500mg, 700mg, 900mg, 1200mg, 1600mg, 2100mg, 2700mg and 3000mg .
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Dose Escalation-Part 1, Expansion-Part 2 (Experimental): In part 1, escalating dose cohort, patients will receive intravenous infusions of EMB-01 weekly (QW). The duration of each treatment cycle is 28 days (4 weeks). Dose escalation will continue until the maximum tolerated dose (MTD) or recommended phase II dose (RP2D) is reached or all planned doses are administered.
  In part 2, participants will receive intravenous infusion of EMB-01 at the recommended Phase II dose (RP2D) regimen(s) once weekly. The duration of each treatment cycle is 28 days (4 weeks).
  Interventions: Drug: EMB-01

INTERVENTIONS:
Drug: EMB-01 — In part 1, patients will receive intravenous infusions of EMB01 weekly (QW). Dose escalation will continue until the maximum tolerated dose (MTD) or recommended phase II dose (RP2D) is reached or all planned doses are administered.
  In part 2, participants will receive intravenous infusion of EMB-01 at RP2D
  The duration of each treatment cycle in both part 1 and part 2 is 28 days (4 weeks).
  Participants may continue to receive study drug until discontinuation criteria are met.
  Other Names: FIT-013a

SUMMARY:
First-in-human, Phase I/II, Multicenter, Open-Label Study of EMB-01 in Patients with Advanced/Metastatic Solid Tumors

DETAILED DESCRIPTION:
This is a first-in-human (FIH), open-label, Phase I/II study of EMB-01, a bispecific Epidermal growth factor receptor (EGFR) and c-Mesenchymal-Epithelial Transition (cMet) antibody, in patients with advanced solid tumors who have progressed on available standard therapies or for which no standard therapy exists. The study consists of two parts: Phase I (dose escalation) and Phase II (cohort expansion). The study is planning to recruit tentatively 33-66 subjects with advanced/metastatic solid tumors in phase I and approximately 42-120 subjects with EGFR mutant and/or cMET aberrated NSCLC who have progressed on or are intolerant to standard treatment(s) (including platinum-based therapy) will be enrolled at the RP2D(s) in phase II part of the study. In phase II, patients will be assigned to five groups according to their molecular status at baseline. The trial will consist of molecular pre-screening period (Phase II only), clinical screening period (-28 to -1 days), treatment cycles (each cycle is 28 days, maximum up to 2 years), and safety follow-up period (30 days after the last dose).

ELIGIBILITY:
Inclusion Criteria:

Molecular Pre-screening Inclusion criteria (Phase II only)

1. The patient must sign the molecular pre-screening Inform Consent to allow for the molecular pre-screening process. All patients must have documented evidence of EGFR and/or cMet aberrations.

Screening Inclusion Criteria

1. Able to understand and willing to sign the Informed Consent Form (ICF).
2. Histologically/cytologically confirmed advanced/metastatic solid tumors with measurable disease [Response Evaluation Criteria in Solid Tumors (RECIST) v1.1]:

   Phase I: advanced/metastatic solid tumors including but not limited to NSCLC, colorectal cancer, gastric cancer and liver cancer refractory to standard therapy or for which no standard therapy is available or accessible.

   Phase II: Advanced/metastatic NSCLC Patients have confirmed EGFR mutant and/or cMET aberration, and have progressed after standard treatment (including platinum-based therapy) or are intolerant to standard treatment. Additionally, patients with T790M mutation have received FDA/Health Authority approved therapies (if accessible) for this indication (i.e., osimertinib) and have progressed or became intolerant.

   A patient who has refused all currently available therapy is allowed to enroll, but must be documented in the source record.
3. Must have adequate organ function.
4. Regarding prior anti-tumor therapy:

   1. Must have stopped treatment at least 4 weeks or within 5 half-lives.
   2. Generalized radiation therapy must have stopped 3 weeks before first dose of EMB 01, or local radiotherapy or radiation therapy for bone metastases must have stopped 2 weeks before first dose of EMB-01. No therapeutic radiopharmaceuticals are taken within 8 weeks before first dose of EMB-01.
   3. Patients must have recovered to ≤Grade 1 from the adverse effects of such above treatment before beginning study treatment.
5. Female patient with fertility or male patient whose partner has fertility should use one or more contraceptive methods for contraception starting from screening period and continue throughout the study treatment and for 3 months.
6. ECOG score 0 or 1 for phase I, and ≤2 for phase II.

Exclusion Criteria:

Molecular Pre-screening Exclusion Criteria (Phase II only)

Subject who meets any of the follow criteria can't be proceeded to clinical screening:

1. Patients who are unwilling to sign the molecular pre-screening ICF.
2. Patients for whom local EGFR and/or cMET data or the results of central laboratory testing do not meet the molecular pre-screening inclusion criteria.

Screening Exclusion Criteria

1. Life expectancy < 3 months.
2. Subject with primacy central nervous system (CNS) malignancy or symptomatic CNS (leptomeningeal or brain) metastases.
3. Pregnant or nursing females.
4. Subjects who have had major surgery within 28 days prior to screening.
5. Serious underlying medical conditions, including but not limited to un-controlled hypertension, other cardiovascular disease or diabetes, ongoing or active infection, psychiatric, psychological, familial or geographical condition that, in the judgment of the investigator, may interfere the compliance with study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 186 (Estimated)
Dates: Start 2018-12-13 (Actual); Primary Completion 2025-03-14 (Estimated); Study Completion 2026-01-15 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) (phase 1 only) | cycle 1 (1cycle = 28 days)
  Maximum tolerated dose
Adverse Events (AEs), and Serious Adverse Events (SAEs) | Screening up to follow-up (30 days after the last dose)
  Adverse Events, and Serious Adverse Events
Overall Response Rate (ORR) (phase 2 only) | From the date fo dosing until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 48 months
  Overall Response Rate

SECONDARY OUTCOMES:
Maximum Serum Concentration (Cmax) | Through treatment discontinuation: an average of 6 months
  Maximum Serum Concentration
Area Under the Plasma Concentration-Time Curve (AUC) | Through treatment discontinuation: an average of 6 months
  Area Under the Plasma Concentration-Time Curve
Trough Serum Concentration (Ctrough) | Through treatment discontinuation: an average of 6 months
  Trough Serum Concentration
Elimination half-life (t1/2) | Through treatment discontinuation: an average of 6 months
  Elimination half-life
Clearance (CL) | Through treatment discontinuation: an average of 6 months
  Clearance
Volume of distribution at steady state (Vss) | Through treatment discontinuation: an average of 6 months
  volume of distribution at steady state
Accumulation Ratio (AR) | hrough treatment discontinuation: an average of 6 months
  Accumulation Ratio
Dose Proportionality | Through treatment discontinuation: an average of 6 months
  Dose Proportionality
Anti-Drug Antibodies (ADA) | Through study completion, an average of 7 months
  Anti-Drug Antibodies
Duration Of Response (DOR) | From the date fo dosing until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 48 months
  Duration Of Response
Progression-Free Survival (PFS) | Through treatment discontinuation: an average of 6 months
  Progression-free survival

OTHER OUTCOMES:
Pharmacodynamic (Soluble EGFR and cMET concentration) | Through treatment discontinuation: an average of 6 months
  Pharmacodynamic (Soluble EGFR and cMET concentration)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (3):
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Gabrail Cancer Center Research, Canton, Ohio
- China (2):
  - Guangdong General Hospital, Guangzhou, Guangdong
  - Shanghai Chest Hosptial, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No